CLINICAL TRIAL: NCT02404181
Title: Validation of a Delirium Monitor in Postoperative Elderly Patients
Brief Title: Validation of a Delirium Monitor
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: University Medical Center Nijmegen (Other); Isala (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, A.J.C. Slooter, MD, PhD, UMC Utrecht
Other Study IDs: NL46622.041.13
Record Dates: First submitted 2015-03-02; First posted 2015-03-31 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Delirium
Keywords: Validation Studies; EEG
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Days
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Delirium is a common disorder in hospitalized patients, nevertheless it is poorly recognized by physicians and nurses, even when screening instruments are used. Electroencephalography (EEG) appears to be a sensitive tool for the diagnosis of delirium. However, standard EEG recording with 25 electrodes is labor intensive. We have previously showed that a brief EEG registration with three electrodes and automatic processing can distinguish patients with delirium from patients without delirium very well. However, these findings need to be validated in an unselected population.

The primary objective of this validation study is to investigate the sensitivity, specificity, and predictive values of the EEG-based delirium monitor (including three electrodes and a reference electrode) compared to delirium quantification in frail elderly patients after surgery.

In an international multicenter study, 154 frail elderly patients will be included who will undergo elective surgery and are expected to remain admitted for at least two postoperative days. Patients are excluded if communication is not possible or admitted for neurological surgery.

A five minute EEG registration with the delirium monitor with four electrodes will be performed prior surgery and three consecutive days after surgery or until discharge. Within one hour of the EEG recording, the delirium assessment will be performed and recorded on video, which will be evaluated by delirium experts. The relative delta power (calculated from one minute of artifact-free EEG segment) will be compared with the conclusion of the delirium experts.

ELIGIBILITY:
Inclusion Criteria:

* 60 years and older
* Frail
* Undergoing elective surgery
* Expected to remain admitted for at least 2 postoperative days

Exclusion Criteria:

* No communication possible due to a language barrier or deafness
* Admission for neurological surgery
* Participation in this study during a previous hospital admission
* Practical or logistical reasons hampering the use of the delirium monitor, such as technical failure of the monitor
* Isolation because of known carrier ship of a resistant bacterium

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source population will consist of frail, elderly patients (≥60 years) who will undergo elective surgery in the University Medical Center Utrecht, Isala Clinics Zwolle, Radboud University Medical Center Nijmegen, or Charité Universitätsmedizin Berlin, and who will be expected to remain admitted for at least two postoperative days. These patients will be informed on this study before admission to the hospital.
Sampling Method: Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2014-03; Primary Completion 2016-07-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Relative delta power (based on 1 min. artifact-free data) will be compared to the classification of the delirium expert in elderly postoperative patients resulting in the sensitivity, specificity and predictive values of the delirium monitor for each day | 4 days

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Numan T, van den Boogaard M, Kamper AM, Rood PJT, Peelen LM, Slooter AJC; Dutch Delirium Detection Study Group. Delirium detection using relative delta power based on 1-minute single-channel EEG: a multicentre study. Br J Anaesth. 2019 Jan;122(1):60-68. doi: 10.1016/j.bja.2018.08.021. Epub 2018 Oct 2. PMID 30579407